CLINICAL TRIAL: NCT07300982
Title: Studies of Insulin and Glucagon Action in the Liver
Acronym: SIGNAL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00117291; R01DK141090 (NIH)
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetes (DM)
Keywords: Glucose metabolism; Hepatic insulin sensitivity; Glucagon; Insulin; hepatic glucose production
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Glucagon; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The studies proposed here will focus on the hepatic interactions of insulin and glucagon using physiological concentrations of these two islet peptides. A group of healthy subjects will be studied on two occasions over 2 weeks in counterbalanced order (with and without glucagon) during a glucose clamp with a fixed dose of insulin. Hepatic glucoses production and glucose metabolism will be measured with stably labeled glucose tracers.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucagon infusion during hyperinsulinemic clamp (Experimental): Glucagon infusion either graded (0.2→0.4→0.6 ng/kg/min) or continuous (0.4 ng/kg/min) during the final 90 minutes of a hyperinsulinemic glucose clamp. The graded or continuous glucagon infusions are given as a component of 2 separate protocols.
  Interventions: Drug: Glucagon
- Saline infusion during hyperinsulinemic clamp (Placebo Comparator): Saline infusion during the final 90 minutes of an otherwise identical clamp procedure.
  Interventions: Drug: Saline (placebo)

INTERVENTIONS:
Drug: Glucagon — Glucagon infusion either graded (0.2→0.4→0.6 ng/kg/min) or continuous (0.4 ng/kg/min) during the final 90 minutes of a hyperinsulinemic glucose clamp. The graded or continuous glucagon infusions are given as a component of 2 separate protocols. Glucagon prepared per pharmacy/bedside protocol.
  Arms: Glucagon infusion during hyperinsulinemic clamp
Drug: Saline (placebo) — IV saline infusion during clamp for 90 minutes as control.
  Arms: Saline infusion during hyperinsulinemic clamp

SUMMARY:
This study examines how glucagon works to regulate glucose metabolism, based on new findings that suggest glucagon signaling in the liver has more than one role, and that these multiple roles can be opposing in nature. Understanding this biology provides an opportunity to develop new generations of glucagon-based drugs that target specific pathways, making them more effective at controlling blood glucose.

Participants will complete paired, 5-hour hyperinsulinemic glucose clamp visits in which they receive either glucagon or saline infusions while blood glucose is maintained and frequent blood samples are collected. The primary focus is whether coordinated glucagon and insulin signaling enhances hepatic insulin sensitivity.

DETAILED DESCRIPTION:
Volunteers will undergo screening for medical history, medication usage, and blood work; those who qualify will be offered participation. Study participation will last approximately 5-12 weeks depending on appointment availability and the number of infusions planned. This protocol involves two sets of paired procedures. Approximately 15 participants will complete each set of paired visits. Participants can opt to complete one set of paired visits or both sets of paired visits.

Set 1: Each participant will complete two 5-hour hyperinsulinemic clamp procedures to examine the effects of glucagon on glucose metabolism while measuring systemic glucose turnover and related blood markers. The procedures will be identical, except for the final phase of the procedure when either saline or a stepwise glucagon infusion will be administered.

Set 2: Each participant will complete two 5-hour hyperinsulinemic clamp procedures to examine the effects of insulin on glucose metabolism while measuring systemic glucose turnover and related blood markers. The procedures will be identical, except for the final phase of the procedure when either saline or a steady glucagon infusion will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 18-45 years
* Body Mass Index (BMI) < 27.0 kg/m²
* Fasting plasma glucose ≤ 95 mg/dL or HbA1c ≤ 5.8% as measured at screening visit

Exclusion Criteria:

* Active medical disease: e.g. active infectious, inflammatory, neurodegenerative or mental health disorders
* No personal history of diabetes or pancreatitis
* No personal history of cardiac, gastrointestinal, renal or liver disease
* No history of diabetes among any first-degree family members
* Renal insufficiency (eGFR < 60 mL/kg/min)
* Anemia (hematocrit < 34%) as measured at screening visit
* Pregnant females
* Consumption of daily medications that alter glucose metabolism of GI function (glucocorticoids, psychotropics, narcotics, metoclopramide)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Glucose appearance (Ra) | In these experiments outcomes will be based on measurements made in the final 90 minutes of the hyperinsulinemic glucose clamp.
  Glucose appearance will be determined using steady state computations, unless a stable tracer:tracee ratio is not maintained
Glucose disappearance (Rd) | In the experiments described here glucose turnover (Ra and Rd) will be determined in the final 90 minutes of the hyperinsulinemic glucose clamp.
  Glucose disappearance (Rd) will be determined using steady state computations, unless a stable tracer:tracee ratio is not maintained
Hepatic insulin sensitivity | Basal period (time -30-0 min), after the insulin infusion alone (60-90 min), and during the glucagon/saline infusions (120-180 min)
  Hepatic insulin sensitivity will be calculated as EGP divided by insulin concentration

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No